CLINICAL TRIAL: NCT07080099
Title: Effects of Bimanual Intensive Therapy With Sensory Training on Motor Function, Sensory Function and Functional Independence in Post Stroke Patients
Brief Title: Effects of Bimanual Intensive Therapy With Sensory Training in Post Stroke Patients
Acronym: BIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0236
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; bimanual intensive training; sensory training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the study would be single blinded as the assessor of the study would be kept blind of the treatment groups to which patients will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bimanual intensive with passive sensory training (Experimental): Group A will receive bimanual intensive therapy with sensory training of 45 minutes with short resting intervals. Treatment will be given 3 times per week for 8 weeks.
  Interventions: Other: BIMANUAL INTENSIVE THERAPY WITH PASSIVE SENSORY TRAINING
- Bimanual intensive with active sensory training (Experimental): Group B will receive bimanual intensive therapy with active sensory training of 45 minutes with short resting interval given to the patient. The treatment will be given 3 times per week for 8 weeks.
  Interventions: Other: BIMANUAL INTENSIVE THERAPY WITH ACTIVE SENSORY TRAINING

INTERVENTIONS:
Other: BIMANUAL INTENSIVE THERAPY WITH PASSIVE SENSORY TRAINING — Bimanual intensive therapy Bimanual coordination training ,Functional training of the hands ,Trask oriented training, Bilateral arm training,
  Passive sensory training:
  Electrical stimulation.
  Arms: Bimanual intensive with passive sensory training
Other: BIMANUAL INTENSIVE THERAPY WITH ACTIVE SENSORY TRAINING — Bimanual intensive therapy:
  * Bimanual coordination training ,Functional training of the hands
  * Trask oriented training, bilateral arm reaching
  Active sensory training:
  sensory re education techniques ,touching different objects, massage, identifying different temperatures, and sensory locating.
  Arms: Bimanual intensive with active sensory training

SUMMARY:
Stroke is the major serious health burden and the leading cause of serious long term disability around the world. One of the most cumbersome deficits after a stroke is impairment in the contralateral upper limb. Bimanual intensive therapy (BIT) is a specialized approach used in rehabilitation for individuals, typically children, who have hemiplegia or hemiparesis, which means weakness or paralysis on one side of the body A therapy strategy known as "sensory training" aims to improve sensory integration and processing in people who struggle with sensory processing issues. The aim of this study is to determine the combined effects of bimanual intensive therapy with sensory training in addition conventional therapy on motor functions, sensory function and functional independence stroke patients.

DETAILED DESCRIPTION:
This randomized clinical trial, will be conducted at jinnah hospital Lahore. For this study, the estimated sample size will be 38. The participants will be randomly allocated using online randomization tool into two groups; group A will receive the bimanual intensive training with passive sensory training for 45 minutes. Group B will receive bimanual intensive training with active sensory training for 45 minutes. Each participants will receive treatment for three days on alternative days for 8 weeks.

Fugal Meyer assessment will be used to asses' motor function. Nottingham Sensory assessment will be used to asses' sensory functions and Functional independence measure for activities of daily living. The data will be entered and analyzed using SPSS 26. Statistical significance will be set at p=0.05. Normality of data will be assessed through kolmogrove-smirnov test and shapirno-wilk test. Assessment will be carried out at bassline, 4th week and 8th week follow-up. For between group analyses of parametric data independent T test will be used, while Man Whitney test will be used for non-parametric data. For within groups comparison repeated measure Annona will be used, for non-parametric, Freidman Annona will be applied

ELIGIBILITY:
Inclusion Criteria:

* Patients with age group 45 to 65
* Both genders
* Patients with stroke that was diagnosed clinically and/ or by computed tomography (CT) or magnetic resonance imaging
* Patient with stable vital signs and GCS score >8-15
* Patients with mini mental state examination score>24(30)

Exclusion Criteria:

* Patients with severe cardiopulmonary complications
* Patients with history of epilepsy
* Patients with the presence of a pacemaker
* Patients with an history of an intracranial implant
* Patients with presence of a cranial defect
* Any other neurological conditions

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
FUGAL MEYER ASSESSMENT (FMA) | 8 weeks
  The FMA assessment contained 33 items (divided into nine domains) regarding different movements, reflexes, and coordination. The assessment includes functional classes of upper extremity reflex activities, flexor synergy motion, extensor synergy motion, activities that were accompanied by synergy motion, disengaging movement, normal reflex action, and carpal joint stability.
NOTTINGHAM SENSORY ASSESSMENT | 8 weeks
  The Nottingham Sensory Assessment is a standardized scale for assessing sensory impairment in stroke patients.
FUNCTIONAL INDEPENDENCE MEASURE (FIM) | 8 weeks
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of a disability of populations. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.

CONTACTS AND LOCATIONS:
Overall Officials: muhammad kashif, PHD, Study Chair — Riphah International University
Locations (1):
- Muhammad kashif, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunner IC, Skouen JS, Strand LI. Is modified constraint-induced movement therapy more effective than bimanual training in improving arm motor function in the subacute phase post stroke? A randomized controlled trial. Clin Rehabil. 2012 Dec;26(12):1078-86. doi: 10.1177/0269215512443138. Epub 2012 May 4. PMID 22561098
- [Background] Ribeiro DKMN, Lenardt MH, Lourenco TM, Betiolli SE, Seima MD, Guimaraes CA. The use of the functional independence measure in elderly. Rev Gaucha Enferm. 2018 Jun 7;38(4):e66496. doi: 10.1590/1983-1447.2017.04.66496. English, Portuguese. PMID 29933424
- [Background] Zamarro-Rodriguez BD, Gomez-Martinez M, Cuesta-Garcia C. Validation of Spanish Erasmus-Modified Nottingham Sensory Assessment Stereognosis Scale in Acquired Brain Damage. Int J Environ Res Public Health. 2021 Nov 29;18(23):12564. doi: 10.3390/ijerph182312564. PMID 34886287
- [Background] Lin SH, Dionne TP. Interventions to Improve Movement and Functional Outcomes in Adult Stroke Rehabilitation: Review and Evidence Summary. J Particip Med. 2018 Jan 18;10(1):e3. doi: 10.2196/jopm.8929. PMID 33052128
- [Background] Arya KN, Pandian S, Agarwal GG, Chaudhary N, Joshi AK. Effect of NEuroplasticity-Principles-based SEnsory-Rehabilitation (NEPSER) on sensori-motor recovery in stroke: study protocol for a randomized controlled trial. Neurol Res Pract. 2021 Feb 4;3(1):8. doi: 10.1186/s42466-021-00108-1. PMID 33536067
- [Background] Huang JJ, Pei YC, Chen YY, Tseng SS, Hung JW. Bilateral Sensorimotor Cortical Communication Modulated by Multiple Hand Training in Stroke Participants: A Single Training Session Pilot Study. Bioengineering (Basel). 2022 Nov 24;9(12):727. doi: 10.3390/bioengineering9120727. PMID 36550934
- [Background] Norwood MF, Lakhani A, Watling DP, Marsh CH, Zeeman H. Efficacy of Multimodal Sensory Therapy in Adult Acquired Brain Injury: A Systematic Review. Neuropsychol Rev. 2023 Dec;33(4):693-713. doi: 10.1007/s11065-022-09560-5. Epub 2022 Sep 2. PMID 36056243
- [Background] Stoykov ME, Heidle C, Kang S, Lodesky L, Maccary LE, Madhavan S. Sensory-Based Priming for Upper Extremity Hemiparesis After Stroke: A Scoping Review. OTJR (Thorofare N J). 2022 Jan;42(1):65-78. doi: 10.1177/15394492211032606. Epub 2021 Jul 26. PMID 34311607
- [Background] Kim KH, Jang SH. Effects of Cognitive Sensory Motor Training on Lower Extremity Muscle Strength and Balance in Post Stroke Patients: A Randomized Controlled Study. Clin Pract. 2021 Sep 14;11(3):640-649. doi: 10.3390/clinpract11030079. PMID 34563008
- [Background] Arya KN, Pandian S, Joshi AK, Chaudhary N, Agarwal GG. Active Sensory Therapies Enhancing Upper Limb Recovery Among Poststroke Subjects: A Systematic Review. Ann Neurosci. 2022 Apr;29(2-3):104-115. doi: 10.1177/09727531221086732. Epub 2022 Apr 3. PMID 36419520
- [Background] Sim TY, Kwon JS. Comparing the effectiveness of bimanual and unimanual mirror therapy in unilateral neglect after stroke: A pilot study. NeuroRehabilitation. 2022;50(1):133-141. doi: 10.3233/NRE-210233. PMID 34957959
- [Background] Stinear CM, Lang CE, Zeiler S, Byblow WD. Advances and challenges in stroke rehabilitation. Lancet Neurol. 2020 Apr;19(4):348-360. doi: 10.1016/S1474-4422(19)30415-6. Epub 2020 Jan 28. PMID 32004440
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] Taylor TN, Davis PH, Torner JC, Holmes J, Meyer JW, Jacobson MF. Lifetime cost of stroke in the United States. Stroke. 1996 Sep;27(9):1459-66. doi: 10.1161/01.str.27.9.1459. PMID 8784113